CLINICAL TRIAL: NCT00013234
Title: Health Services Implications of a Teledermatology Consult System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IIR 98-159
Record Dates: First submitted 2001-03-14; First posted 2001-03-16 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2007-02

CONDITIONS: Teledermatology

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Other)
  Interventions: Procedure: Teledermatology

INTERVENTIONS:
Procedure: Teledermatology

SUMMARY:
We have previously shown (IIR 95-045) that teledermatology, using store and forward technology, can result in reliable and accurate diagnostic outcomes when compared to clinic-based dermatology consultations. This investigation builds on that fundamental diagnostic information by assessing the health services implications of a teledermatology consult system.

DETAILED DESCRIPTION:
Background:

We have previously shown (IIR 95-045) that teledermatology, using store and forward technology, can result in reliable and accurate diagnostic outcomes when compared to clinic-based dermatology consultations. This investigation builds on that fundamental diagnostic information by assessing the health services implications of a teledermatology consult system.

Objectives:

To investigate health services outcomes related to teledermatology implementation. Outcomes of interest were time to diagnosis and treatment initiation, the proportion of patients that avoided the need for a clinic-based encounter, and an economic analysis.

Methods:

Patients referred from the primary care clinics to the dermatology consult service were randomized to either usual care or a teledermatology consultation. A usual care consultation consisted a conventional text-based electronic consult request. A teledermatology consultation included digital images and a standardized history, in addition to the electronic text-based consult. Consultant dermatologists, reviewing the consult requests for both modalities, decided when, and if, a referral required a clinic-based evaluation.

Status:

Final report has been prepared and is in the review process at this time.

ELIGIBILITY:
Inclusion Criteria:

Patients referred to Dermatology Consult Service.

Exclusion Criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Study Completion 2003-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John D. Whited, MD MHS, Principal Investigator — Durham VA Medical Center, Durham, NC; Eugene Z. Oddone, MD MHSc, Principal Investigator — Durham VA Medical Center, Durham, NC
Locations (1):
- Durham VA Medical Center, Durham, NC, Durham, North Carolina, United States

REFERENCES:
- [Result] Whited JD, Datta S, Hall RP, Foy ME, Marbrey LE, Grambow SC, Dudley TK, Simel DL, Oddone EZ. An economic analysis of a store and forward teledermatology consult system. Telemed J E Health. 2003 Winter;9(4):351-60. doi: 10.1089/153056203772744671. PMID 14980092
- [Result] Whited JD. Teledermatology research review. Int J Dermatol. 2006 Mar;45(3):220-9. doi: 10.1111/j.1365-4632.2004.02427.x. PMID 16533219
- [Result] Whited JD, Hall RP, Foy ME, Marbrey LE, Grambow SC, Dudley TK, Datta SK, Simel DL, Oddone EZ. Patient and clinician satisfaction with a store-and-forward teledermatology consult system. Telemed J E Health. 2004 Winter;10(4):422-31. doi: 10.1089/tmj.2004.10.422. PMID 15689645
- [Result] Whited JD. The quality of telemedicine research. J Telemed Telecare. 2006;12(6):271-3. doi: 10.1258/135763306778558114. No abstract available. PMID 17022832
- [Result] Whited JD. Teledermatology. Current status and future directions. Am J Clin Dermatol. 2001;2(2):59-64. doi: 10.2165/00128071-200102020-00001. PMID 11705304
- [Result] Whited JD, Hall RP, Foy ME, Marbrey LE, Grambow SC, Dudley TK, Datta S, Simel DL, Oddone EZ. Teledermatology's impact on time to intervention among referrals to a dermatology consult service. Telemed J E Health. 2002 Fall;8(3):313-21. doi: 10.1089/15305620260353207. PMID 12419025